CLINICAL TRIAL: NCT03711240
Title: Study to Investigate Efficacy of Bevacizumab Combined With Modified-FOLFOXIRI in Patients With Borderline Resectable Colorectal Liver Metastases
Brief Title: The Efficacy of Bevacizumab Combined With m-FOLFOXIRI in Borderline Resectable Colorectal Liver Metastases
Acronym: CBL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-10
Record Dates: First submitted 2018-10-12; First posted 2018-10-18 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer
Keywords: colorectal liver metastases; FOLFOXIRI; bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bevacizumab+mFOLFOXIRI (Experimental)
  Interventions: Drug: bevacizumab; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-FU

INTERVENTIONS:
Drug: bevacizumab — 5mg/kg iv day 1 every 2 weeks
Drug: Oxaliplatin — 85mg/m2 2-hour iv infusion, day 1 every 2 weeks
Drug: Irinotecan — 150mg/m2 1.5-hour iv infusion, day 1 every 2 weeks
Drug: Leucovorin — 200mg/m2 2-hour iv infusion, day 1 every 2 weeks
Drug: 5-FU — 2400mg/m2 46-hour continuous iv infusion, day 1 every 2 weeks

SUMMARY:
This single-arm study will evaluate the resection rate of liver metastases in patients with metastatic colorectal cancer and borderline unresectable liver metastases receiving treatment with bevacizumab in combination with modified-FOLFOXIRI as first line treatment. Patients will receive bevacizumab (5 mg/kg) plus modified-FOLFOXIRI (irinotecan 150 mg/m2, oxaliplatin 85 mg/m2, leucovorin 200 mg/m2, and fluorouracil 2400 mg/m2 as a 46-h continuous infusion) every 14 days as neoadjuvant chemotherapy regimen. This study treatment will continue until surgery, disease progression, unacceptable toxicity, or patient refusal.

DETAILED DESCRIPTION:
This is a phase II study to investigate the efficacy of biweekly bevacizumab in combination with modified-FOLFOXIRI regimen, as first-line chemotherapy in patients with borderline resectable colorectal liver metastases. Borderline resectable liver metastases are considered to have poor-risk diseases infeasible for upfront resection, but own the potential for resection after down-staging. The primary purpose of the study is to determine the resection rate of liver metastases in patients receiving this combination regimen. The secondary objectives are to determine the response rate, progression free survival, overall survival, and safety profiles.

Eligible patients will receive a triplet chemotherapy consisting of bevacizumab (5 mg/kg) plus modified-FOLFOXIRI (irinotecan 150 mg/m2, oxaliplatin 85 mg/m2, leucovorin 200 mg/m2, and fluorouracil 2400 mg/m2 as a 46-h continuous infusion) every 14 days as a cycle. Resectability of primary tumor and liver metastases will be assessed after five cycles of combination treatment with feasible image exams. Patients with progressive disease will be discontinued in this study. For patients feasible for tumor resection, the modified triplet chemotherapy without bevacizumab combination will be continued for one other cycle for patients before surgery. If patients don't reach both the feasibility of tumor resection and progressive disease, another four cycles of bevacizumab combined with modified-FOLFOXIRI could be continued by investigator's judgement. Reassessment of resectability for primary tumor and liver metastases will be conducted using feasible image exams after a total of 9 cycles of combination treatment in these patients. Similarly, the triplet chemotherapy without bevacizumab combination will be continued for the other one cycle before surgery for these patients feasible for tumor resection after reassessment. Bevacizumab should be stopped at least 4 weeks before the planned day of surgery. Short-course radiotherapy will be allowed before surgery for patients with rectal cancer. All patients will be discontinued in this study after tumor resection. Treatment will also be discontinued if the patient requests or the investigator decides that therapy should be withdrawn. Further tumor treatment after treatment discontinuation will be decided based on investigator's judgement with the best knowledge.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of colorectal cancer.
2. Borderline resectable liver metastases of colorectal cancer considered to have poor-risk disease not deemed to be suitable for upfront resection if they had one or more of the following features assessed by a local multidisciplinary team: more than four metastases, any liver lesion with diameter >5 cm, location and distribution of metastatic disease within the liver unsuitable for resection with clear margins (e.g. involvement of both lobes of liver, invasion of intrahepatic vascular structures), extent of liver involvement precluding resection with adequate post-resection residual liver parenchyma volume for viable liver function in the immediate postoperative period, and inability to retain adequate vascular inflow and outflow to maintain viable liver function.
3. At least one measurable lesion according to RECIST criteria.
4. Age 20-75 years.
5. ECOG performance < 1 if age < 70 years, ECOG PS = 0 if age = 70-75 years.
6. Life expectancy of at least 12 weeks.
7. Neutrophils ≥1.5 x 109/L, Platelets≥ 100 x 109/L, Hgb ≥10 g/dl.
8. Total bilirubin ≤1.5 time the upper-normal limits (UNL) of the Institutional normal values and ASAT (SGOT) and/or ALAT (SGPT) ≤5 x UNL, alkaline phosphatase ≤5 x UNL.
9. Serum creatinine≤ 1.5 x UNL.
10. Patients discovered to have proteinuria on urinalysis at baseline, should undergo a 24-hour urine collection and must demonstrate ≤1 g of protein/24 hr.
11. Written informed consent.

Exclusion Criteria:

1. Prior neoadjuvant or adjuvant chemotherapy completed <6 months.
2. Prior chemotherapy for metastatic disease.
3. Any extrahepatic metastases.
4. History or evidence upon physical examination of CNS disease unless adequately treated (e.g., seizure not controlled with standard medical therapy or history of stroke).
5. Serious, non-healing wound, ulcer, or bone fracture.
6. Evidence of bleeding diathesis or coagulopathy.
7. Uncontrolled hypertension.
8. Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤ 6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication.
9. Current or recent (within 10 days prior to study treatment start) ongoing treatment with anticoagulants for therapeutic purposes.
10. Chronic daily treatment with aspirin .
11. Patients with known allergy to Chinese hamster ovary cell proteins, or any of the components of the study medications.
12. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of sin basal cell carcinoma or cervical cancer in situ.
13. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study.
14. Other severe systemic diseases without stable medical control.
15. Pregnant or lactating women.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Resection rate of liver metastases | 6 months
  The percentage of the number of subjects with R0 and R1 resection after treatment.

SECONDARY OUTCOMES:
Tumor response rate | 6 months
  The percentage of the number of subjects with tumor response after combination treatment evaluated using the RECIST criteria version 1.1.
Progression free survival | 5 years
  Time duration measured from the day of registration until the first observation of disease progression based on image exam findings or investigator clinical judgement.
Overall survival | 5 years
  Time duration between the day of registration and the date of death or the last date the patient was known to be alive.
Percentage of adverse effects related to combination treatment | 5 years
  The percentage of subjects with adverse effects related to combination treatment evaluated using the CTCAE criteria version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Shang Hung Chen, Principal Investigator — National Health Research Institutes, Taiwan
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No